CLINICAL TRIAL: NCT04314063
Title: Knowledge,Attitude and Practice of Food Handleres About Food Safety in Assiut University Hospitals
Brief Title: Knowledge,Attitude and Practice of Food Handleres About Food Safety
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amarat Mohamed Mahmoud, principal investigator, Assiut University
Other Study IDs: food safety in hospitals
Record Dates: First submitted 2020-03-13; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Food Borne Diseases
MeSH Terms: conditions — Foodborne Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: nasal swap — nasal swap to detect prevalence of staph aureus in food handlers
  Other Names: no other name

SUMMARY:
The heavy burden of food borne diseases causes substantial economic losses to individual , households, health systems and entire nations.

As poor food hygienic practices could contribute food -borne diseases in hospital, so food handlers' knowledge, attitude and practicing is an important factor that is essential in order to lower food borne disease. All three traits; knowledge, attitude and education are compulsory to enable safe food handling practices

DETAILED DESCRIPTION:
Food is vital for life but can only serve such an important purpose if it is safe and secure to ingest . According to Food and Agricultural Organization (FAO), Food safety is defined as" an assurance that food will not cause harm to consumers when it is prepared and/or eaten according to its intended use" .

Food safety is one of food handler responsibilities . Food handler is defined as "any person who directly handles packaged or unpackaged food ,food equipment and utensils, or food contact surfaces and therefore expected to comply with food hygiene requirements".

Food handling includes all steps of storing, processing, preparing, serving, and preserving food until reaching final consumption . The World Health Organization (WHO) also determined five factors connected to the occurrence of food related llnesses including: unhygienic practices and insufficient sanitation by food handlers, inadequate cooking procedures, improper storage without considering temperature requirements, cross contamination, and sourcing food from unsafe places. Most of these factors are under the responsibility of food handlers who are involved in food production and preparation . According to WHO (2015), food borne diarrheal disease kills about two million people yearly, particularly in developing countries . Statistics of Food Safety Conference in 2013 revealed that 30 million Egyptians are infected with dangerous diseases due to contamination of water, food and environment. This made Egypt one of the greatest affected countries by food-borne diseases. The heavy burden of food borne diseases imposes substantial economic losses to individual, households, health systems and entire nations .

As poor food hygienic practices could contribute food -borne diseases in hospital, so food handlers' knowledge, attitude and practicing is an important factor that is essential in order to lower food borne disease. All three traits; knowledge, attitude and education are compulsory to enable safe food handling practices.

This was supported by previous studies that have demonstrated the essential role of inadequate food handling knowledge, attitude and practice in occurrence of food poisoning .

A lot of previous studies worldwide, documented high levels of knowledge, attitude and practice of food safety among food handlers, as in Saudi Arabia, a study was done in 10 hospitals in Madina, illustrated that food service had good food safety knowledge, 77.9% recorded right answers for knowledge of cross contamination and 52.8% recorded right answers for knowledge of food poisoning, and 49.7% gave right answers knowledge of food storage this was accompanied by highly good food safety practices ; 92.6% had good practice . As well as, another study in Jordan, showed that the means of the percentage scores for the knowledge, attitude, practice, were 84.82, 88.88, 89.43, respectively . Another Indonesian study done in teaching hospital and another non-teaching hospital showed that more than 80% of food handlers have good knowledge in safe food handling procedures, good attitude (66%) and good practices (90%). On the other side, an Indian study was done in tertiary hospital, showed that food handlers had poor knowledge of food borne diseases in terms of etiology (46.67%), mode of transmission (33.33%) and mode of prevention (36.67%) with poor attitude(56.67%) that was reflected on practices that affect negatively on food safety . In Egypt, two previous studies illustrated lower knowledge, attitude and practicing among food handlers, for instance; first study done in Sohage Governorate showed that only 39 % of participants had good knowledge, 61.2 % had positive attitudes and 56.3% reported good food safety practice. The second one was done in Ismailia city hospital, only 33.3% of them were aware of the importance of washing hands after handling raw meat. Moreover, 59.1% of them were ignore why raw foods must be kept separate from cooked foods and 64.4% also were unaware of the proper temperature of cooking chicken and only 40.9 % of them were always washing their hands before handling food, in addition , only 27.3% of them were properly clean, sanitize and store equipment.. About 97% of all studied participants need for more information about food safety in the future . However, another study in the kitchens of Ain Shams University Hospitals showed better knowledge and practice; mean knowledge score was 76.6 ± 19.6 and the mean practice score was 68.1 ± 22.4 . Food handlers play a major role in transmitting pathogens passively from contaminated sources such as transmitting pathogens from raw meat to a ready to eat food. They may also carry some human specific food- borne pathogens such as Hepatitis A, Salmonella, Staphylococcus aureus and Shigella sp in their hands, cuts or sores, mouth, skin and hair. In addition, they may also shed food borne pathogens, such as E. coli and Salmonella during the infectious period or less important during recovery period of a gastrointestinal sickness ..

Outbreaks of foodborne infections in hospitals are facilitated by several factors; these include staff carriers, poor hygiene conditions in the kitchens, carelessness and lack of training of food handlers, but all causes are mostly preventable.

So food-services staff in hospitals represents a potential source of nosocomial foodborne outbreaks, since they may possibly introduce pathogens into foods during every phase from purchase to distribution .Food handlers who were S. aureus carrier and have direct contact with prepared food can contaminate pathologic organism to hospital inpatients . It was mentioned that S. aureus colonization rates in the general population were estimated to be approximately 20% - 32%. Regarding studies specific for food handlers, prevalence rates vary among countries. It ranged from 2% of food handlers in a study done in Italy , 12% in Finland, .5% in Ethiopia , 19% in Chile ,57.5% in Botswana and 62% in India . However, another study in the kitchen of Ain shams university hospitals showed 41 % of participants had positive nail swabs likely, another study in Egypt had a similar infection rate with staph aureus (38%) .

ELIGIBILITY:
Inclusion Criteria:

- any person work in nutrition unit

Exclusion Criteria:

* no exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Assiut University Hospitals. Nutrition unit (350)worker. Single large kitchen which is located in ground floor in women health hospital consisting of 4 main sectors according to serving area ( private sector , free patient service, doctors and agriculture unit) (132 )worker.
  Main distribution office for distribution in all Assiut university hospitals peripheral distribution offices (61)worker.
  peripheral distribution units in the following hospitals (105) (neurology, urology, cardiology, pediatric , Tropical and gynecology) 5 hostels (2 in side and 3 outside) (52)worker.
Sampling Method: Probability Sample
Enrollment: 276 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Knowledge, attitude and practices of food handlers about food safety | one year
  A questionnaire was prepared based on validated questionnaires of previous studies Food safety attitudes and self-reported practices were evaluated by a5 level Likert scale.
  For items under the attitudes section, positively worded questions were scored as follows: strongly agree (4), agree (3), neutral (2), disagree (1) and strongly disagree (0). In contra st, for negatively worded items, the lowest point (0) was given to "strongly agree" and the highest (4) for "strongly disagree". The scores given ranged 0-60.
  For positively worded selfreported practices, "always" was scored (4) and the lowest point (0) was given to "never"; this was reversed for the negatively worded questions and the score range was 0-76.
  Total scores equal to or greater than 50% of the maximum scores of knowledge, atti -tude or practice were categorized as "good" while lower scores were considered "poor" or unsatisfactory .

SECONDARY OUTCOMES:
prevalence of staph aureus in food hand handlers | one year
  carrier or non carrier of staph aureus

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Roushdy, MD, Study Director — Assiut University
Locations (1):
- Amarat Mohamed Mahmoud, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dudeja P, Singh A, Sahni N, Kaur S, Goel S. Effectiveness of an intervention package on knowledge, attitude, and practices of food handlers in a tertiary care hospital of north India: A before and after comparison study. Med J Armed Forces India. 2017 Jan;73(1):49-53. doi: 10.1016/j.mjafi.2016.10.002. Epub 2016 Nov 30. PMID 28123245
- [Background] El Derea H, Salem E, Fawzi M, Abdel Azeem M. Safety of patient meals in 2 hospitals in Alexandria, Egypt before and after training of food handlers. East Mediterr Health J. 2008 Jul-Aug;14(4):941-52. PMID 19166178
- [Background] Buccheri C, Casuccio A, Giammanco S, Giammanco M, La Guardia M, Mammina C. Food safety in hospital: knowledge, attitudes and practices of nursing staff of two hospitals in Sicily, Italy. BMC Health Serv Res. 2007 Apr 3;7:45. doi: 10.1186/1472-6963-7-45. PMID 17407582